CLINICAL TRIAL: NCT06898827
Title: Distraction Therapy Using Virtual Reality in Patients Undergoing Cardiac Rehabilitation: Effects on Cardiac Efficiency, Anxiety and Exercise Tolerance
Brief Title: Distraction Therapy Using Virtual Reality in Cardiac Rehabilitation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Anabel Sciriha, Principal Investigator, University of Malta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Cardiac Rehab & VR
Record Dates: First submitted 2025-01-22; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Disease; Coronary Artery Bypass
Keywords: Cardiac Rehabilitation; Virtual Reality; Rehabilitation
MeSH Terms: conditions — Heart Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A minimum of 20 patients undergoing phase 3 of CR shall be recruited in this study. All patients who are suffering from any cardiac condition or have had a cardiac event and are referred for cardiac rehabilitation are eligible to participate. Patients with Atrial Fibrillation, those with an implantable cardioverter defibrillator or a pacemaker and any patients known to suffer from Vertigo shall be excluded from the study. Those patients showing an interest in participating shall be offered information about what the study entails by the intermediary, this being the cardiac rehabilitation nurse. Upon consenting, general baseline demographic data including age, weight, height, body mass index (BMI), gender and drug history will be collected. The participants shall then be randomly assigned into two groups being: the control group who shall receive the usual CR programme without the addition of VR, and the intervention group who shall be subject to 20 minutes of IVR2
Who Masked: Investigator
Masking Description: The investigators will be blinded to all participants and their allocated group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The intervention group who shall be subject to 20 minutes of IVR using the MORPHEUS programme, software developed by the Faculty of Information and Technology, when carrying out cycle ergometry during the 6 - week, bi-weekly CR programme. These patients shall carry out 10 minutes of warm up by cycling without IVR, followed by 20 minutes of cycling while wearing the headset with IVR input, followed by another 10 minutes of cool down without IVR input. The duration of 20 minutes input time was based on recommendations set by the Department of Business, Energy and Industrial Strategy, UK (2020) to prevent motion sickness.
  Interventions: Procedure: IVR using the Morpheus Programme; Procedure: Cardiac Rehabilitation control group
- Control (No Intervention): no treatment using VR

INTERVENTIONS:
Procedure: IVR using the Morpheus Programme — Patients in the intervention group will receive 20 mins of immersive therapy during cardiac rehabilitation
  Other Names: IVR
  Arms: Experimental
Procedure: Cardiac Rehabilitation control group — Cardiac rehabilitation but no IVR
  Other Names: Exercise
  Arms: Experimental

SUMMARY:
The European Society of Cardiology has been putting forward the need for new adjuncts or models that optimise outcomes from CR programmes. Immersive virtual reality (IVR) is one of the newest technologies whose input in CR is currently being investigated. It is a technology which helps simulate the real environment through a virtual one, allowing for interaction with the environment and to carry out exercise with variability, where intensity, repetition and feedback are key elements. It is reported that immersion in VR environments diverts the attention of the patient from unpleasant bodily sensations, thus delaying the onset of boredom and fatigue. This is reported to possibly incite higher participation. In addition, VR has some noticeable indirect benefits for postcardiac event patients. It is reported that when using head-mounted devices during stationary cycling, a reduction in sympathetic tone and thus increase blood flow to the muscles prolonging the exercise duration and enhancing fatigue resistance will result. The use of distraction therapy through VR, one which isolates the patients from the medical context and puts all the attention on the virtual experience, makes the patient be distracted from the unpleasant stimuli of the surrounding environment. Distraction therapy through VR is reported to provide positive emotions, reduce anxiety and lead to an underestimation of the treatment duration.

DETAILED DESCRIPTION:
Cardiovascular disease is a leading cause of death and morbidity worldwide, with the WHO reporting 17.9 million of all global deaths in 2019 attributed to cardiovascular disease, with 7.4 million deaths attributed to coronary heart disease. In Europe, CVDs are estimated to cause close to 4 million deaths annually, generating a cost of 196 billion Euros/year. Cardiac rehabilitation, an intervention offered to the majority of patients who would have experience any cardiac event, includes several components delivered by a multi-disciplinary team. The components include health education, advice on cardiovascular risk reduction, physical activity, and stress management. Evidence that cardiac rehabilitation reduces mortality, morbidity, unplanned hospital admissions in addition to improvements in exercise capacity, quality of life and psychological well-being is increasing, and it is now recommended in international guidelines, ones which include the American Heart Association and the American Association of Cardiovascular and Pulmonary Rehabilitation, The Canadian Association of Cardiac Rehabilitation, The European Association of Cardiovascular Prevention and Rehabilitation, The Australian Cardiovascular Health and Rehabilitation Association and The World Health Organization Expert Committee on Rehabilitation after Cardiovascular Diseases. Despite evidence proving all the benefits mentioned above, participation in such interventions is still considered low, and those that complete the programme fail to adhere to exercise after.

The main factors attributing to lack of completion or adherence to CR are depression and anxiety, factors which have been reported to have detrimental effects on self-management behaviours in patients after cardiac surgery. Anxiety has been reported to be independently associated with an increased mortality rate in patients diagnosed with coronary artery disease, particularly in the presence of comorbid depression. Together with this, baseline depression has been associated with the development of a sedentary lifestyle in the long term, as well as with adverse cardiovascular outcomes and increased health care costs. It was reported that depression and anxiety are likely to persist despite cardiac treatment and rehabilitation and if these are not addressed, the positive effects of expensive specialist cardiac procedures and rehabilitation can be diminished. Therefore, the need to determine efficient methods for managing depression and anxiety and improve the outcomes of CR is required.

The European Society of Cardiology has been putting forward the need for new adjuncts or models that optimise outcomes from CR programmes. Immersive virtual reality (IVR) is one of the newest technologies whose input in CR is currently being investigated. It is a technology which helps simulate the real environment through a virtual one, allowing for interaction with the environment and to carry out exercise with variability, where intensity, repetition and feedback are key elements. Immersion in VR environments diverts the attention of the patient from unpleasant bodily sensations, thus delaying the onset of boredom and fatigue. This is reported to possibly incite higher participation. In addition, VR has some noticeable indirect benefits for postcardiac event patients. When using head-mounted devices during stationary cycling, a reduction in sympathetic tone and thus increase blood flow to the muscles prolonging the exercise duration and enhancing fatigue resistance will result. The use of distraction therapy through VR, one which isolates the patients from the medical context and puts all the attention on the virtual experience, makes the patient be distracted from the unpleasant stimuli of the surrounding environment. Distraction therapy through VR is reported to provide positive emotions, reduce anxiety and lead to an underestimation of the treatment duration.

However, although IVR has captured the attention of professionals working in the field of CR, studies in this field are still limited and published protocols are very heterogeneous. IVR has been reported to increase functional capacity, motivation and adherence of patients undergoing CR programmes, however, there is no consensus regarding the outcome measures to be studied, the number of sessions, the protocol to be followed or the technology to be used, since there is great heterogeneity in the scientific literature. Therefore, despite the potential usefulness of the use of VR, there is a need to determine the main short- and medium-term outcome measures in CR programmes.

This research shall therefore investigate whether the inclusion of IVR in patients undergoing phase 3 of CR helps improve anxiety and depression scores, which in turn will increase exercise tolerance and cardiac efficiency when compared to patients who do not have access to this modality.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are suffering from any cardiac condition
* Patients who have had a cardiac event
* Patients referred for cardiac rehabilitation.

Exclusion Criteria:

* Patients with Atrial Fibrillation
* Patients with an implantable cardioverter defibrillator
* Patients with a pacemaker and
* Patients who suffer from Vertigo

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | Up to 6weeks
  Exercise Tolerance test
Hospital Anxiety and Depression Score | Up to 6weeks
  Measure for Anxiety and Depression

CONTACTS AND LOCATIONS:
Overall Officials: Dr Anabel Sciriha, PhD, Principal Investigator — University of Malta; Dr Stephen Lungaro-Mifsud, PhD, Principal Investigator — University of Malta; Dr Tonio Agius, PhD, Principal Investigator — University of Malta
Locations (1):
- Department of Physiotherapy Faculty of Health Sciences, Msida, Malta

IPD SHARING:
Plan to Share IPD: Yes
All information will be coded so each participant information is still anonymous
Supporting Information: Study Protocol, SAP, ICF
Time Frame: September 2024 to June 2025
Access Criteria: The main researchers